CLINICAL TRIAL: NCT02319850
Title: Revisiting the Sarcopenia Diagnosis: New Approaches to Rapid Screening and Preventative Healthcare
Brief Title: Muscle Ultrasound for Sarcopenia Leading to Early Detection
Acronym: MUSCLED
Status: Completed | Type: Observational
Sponsor: George Washington University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); Children's National Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 081320; UL1TR000075 (NIH)
Record Dates: First submitted 2014-12-15; First posted 2014-12-18 (Estimated); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Sarcopenia
Keywords: sarcopenia; screening; geriatrics; muscle; aging; ultrasound
MeSH Terms: conditions — Sarcopenia | interventions — X-Rays

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Reference Group: 18 - 29 years of age; apparently healthy younger participants; 1:1 male and female recruitment ratio (Exposure include DXA scanning).
  Interventions: Radiation: DXA scanning
- Comparison Group: 55 - 75 years of age; apparently healthy older participants; 1:1 male and female recruitment ratio (Exposure include DXA scanning).
  Interventions: Radiation: DXA scanning

INTERVENTIONS:
Radiation: DXA scanning — Exposure: Participants will undergo DXA scanning in the supine position per manufacturer guidelines to estimate absolute and percentage of total lean body mass (LBM) and body fat (BF).
  Other Names: Radiograph, x-rays

SUMMARY:
Sarcopenia is an age-related loss of muscle mass that may affect over 25% of individuals over the age of 60 and results in a 3 to 4 times increased likelihood of developing a disability. Despite these observations, sarcopenia is rarely subject to a systematic screening process as a part of customary geriatric care. Furthermore, when lean body mass (LBM) is measured via dual energy X-ray absorptiometry (DXA) in older adults, it is typically within a reactive, hospital-based, model of healthcare where muscle wasting is only assessed after a loss of functional independence. The investigators propose an affordable, portable screening method with ultrasound imaging to be performed in primary care settings.

The investigators long term goal is to identify individuals at risk, and intervene with treatments that may prevent the onset of debilitating loss of muscle function in the elderly.

DETAILED DESCRIPTION:
Purpose: The overall goal of this pilot project is to validate a rapid, portable, cost-effective, sarcopenia identification method using diagnostic sonography. This method would be used for screening to aid early detection, diagnosis in clinical settings, and monitoring the effects of formal intervention. The investigators central hypothesis is that the sonographic muscle characteristics will be significantly associated with estimates of lean body mass (LBM) and functional status.

Research Setting: George Washington University, Exercise Science Laboratory.

Participants: Subjects will include a healthy young reference group (18 - 29 years of age) and an older comparison group (55 - 75 years of age; n = 15 per group; approximately 50% female), consecutively recruited from George Washington University and the surrounding community.

Implications/Significance: Diagnostic musculoskeletal ultrasound is a portable, inexpensive modality suitable for bedside use or community health initiatives, and features no exposure to low-dose radiation. It is important to note that DXA is considered a relatively low cost procedure, and DXA-based measures may continue to be used as the standard for the sarcopenia syndrome LBM criterion. Consequently, this study will examine if LBM values obtained with ultrasound may serve as a viable proxy of LBM measures obtained with DXA.

The innovation in the investigators study is reflected by a proactive approach to sarcopenia screening that is responsive to the growing shift of healthcare from hospitals to alternative, community-based settings.

ELIGIBILITY:
Inclusion Criteria: You are eligible to participate if:

1. You are between the ages of 18 - 29 years, or 55 - 75 years.
2. You must be able to stand comfortably for 10 minutes and walk a short distance (use of assistive devices are acceptable).

Exclusion Criteria: You are not eligible to participate if:

1. You have a medical condition that results in edema.
2. You have had an upper or a lower extremity amputation.
3. You are, or may be, pregnant.
4. You have a body mass index (BMI) > 30.0.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Enrolled subjects in this pilot study will include a healthy young reference group (18 - 29 years of age) and an older comparison group (55 - 75 years of age; n = 15 per group; approximately 50% female), consecutively recruited from George Washington University and the surrounding community.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2014-02; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sonographic Lean Body Mass | 1 day
  US estimates of aggregate regional LBM (muscle thickness, cm), will be assessed using B-mode diagnostic US with a 13-6 megahertz linear array transducer for morphology measures at 5 axial and appendicular sites.

SECONDARY OUTCOMES:
DXA lean body mass | 1 day
  Participants will undergo dual energy X-ray absorptiometry (DXA) scanning in the supine position per manufacturer guidelines to estimate absolute and percentage of total LBM, and body fat percentage (BF%).
Grip strength | 1 day
  Grip strength will be assessed bilaterally using a isometric dynamometer.
Lower extremity function | 1 day
  A standardized timed sit-to-stand test will be conducted (5 repetitions).
Physical activity questionnaire | 1 day
  Participants will also complete the International Physical Activity Questionnaire (IPAQ) to obtain an estimate of their customary activity and formal exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Loretta DiPietro, PhD, MPH, Principal Investigator — George Washington University
Locations (1):
- George Washington University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Background] Harris-Love MO, Monfaredi R, Ismail C, Blackman MR, Cleary K. Quantitative ultrasound: measurement considerations for the assessment of muscular dystrophy and sarcopenia. Front Aging Neurosci. 2014 Jul 14;6:172. doi: 10.3389/fnagi.2014.00172. eCollection 2014. No abstract available. PMID 25071570